CLINICAL TRIAL: NCT00539513
Title: A Double-Blind Study of N-Acetylcysteine Augmentation in Serotonin Reuptake Inhibitor-Refractory Obsessive-Compulsive Disorder and Depression
Brief Title: N-Acetylcysteine Augmentation in Treatment-Refractory Obsessive-Compulsive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Researchers terminated study due to limited enrollment.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0603001215
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; OCD; glutamate; N-Acetylcysteine; augmentation
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-Acetylcysteine (Experimental): Patients randomized to this arm will receive N-Acetylcysteine augmentation, at a standard dose titrated to 3000 mg within the first week, in addition to the medication regimen they are on at enrollment
  Interventions: Drug: N-Acetylcysteine
- placebo (Placebo Comparator): Patients randomized to this arm will receive placebo, formulated to be indistinguishable from N-Acetylcysteine, in addition to the medication regimen they are on at study enrollment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — 3000 mg by mouth PO (1200 mg AM, 1800 mg PM), 12 weeks
  Other Names: NAC
  Arms: N-Acetylcysteine
Drug: placebo — placebo, 2 capsules PO AM, 3 capsules PO PM, 12 weeks
  Arms: placebo

SUMMARY:
Obsessive-compulsive disorder (OCD) affects 2-3% of the population and leads to a great deal of suffering. Many patients benefit from established treatments, the mainstay of which are cognitive behavioral therapy and a group of antidepressant medications known as serotonin reuptake inhibitors. However, 20-30% of patients get minimal benefit from these established therapeutic strategies. New avenues of treatment are urgently needed.

Existing medications for obsessive-compulsive disorder affect the neurotransmitters serotonin or dopamine; but increasing evidence suggests that functional disruptions of a different neurotransmitter, glutamate, may contribute to some cases of OCD. The researchers are therefore interested in using medications that target glutamate as novel treatment options for those OCD patients who do not benefit from established treatments.

One such medication is the drug N-Acetylcysteine, whose glutamatergic antagonistic properties may be effective in reducing the glutamatergic hyperactivity that is thought to contribute to the pathophysiology of OCD and major depressive disorder (MDD).

Riluzole, which is FDA approved for amyotrophic lateral sclerosis (ALS, or Lou Gehrig's disease) is also a glutamatergic agent. There is evidence that riluzole possesses anti-depressant, anti-obsessional, and anti-anxiety properties.

The modulation of glutamatergic activity is a promising new approach to the treatment of mood disorders. The researchers are therefore now recruiting patients to participate in a double-blind, placebo-controlled trial of N-Acetylcysteine, added to whatever other OCD medications they are taking.

DETAILED DESCRIPTION:
Due to limited participation, this study has closed.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of OCD, confirmed by SCID-IV; symptoms of at least 1 year duration
* moderate to severe OCD symptoms (Y-BOCS > 16)
* documented failure of an adequate trial of an SSRI
* agreement to engage in a reliable form of birth control (women only)

Exclusion Criteria:

* primary diagnosis of a psychotic disorder
* active substance abuse or dependence
* unstable medical condition
* prior exposure to N-Acetylcysteine
* prior psychosurgery
* pregnancy, breastfeeding, or intent to become pregnant during study
* liver function tests (LFTs) elevated to more than 2x the upper limit of normal
* evidence of active liver disease
* seizure disorder
* active suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Pittenger, MD, Ph.D., Principal Investigator — Yale University

REFERENCES:
- [Background] Pittenger C, Krystal JH, Coric V. Glutamate-modulating drugs as novel pharmacotherapeutic agents in the treatment of obsessive-compulsive disorder. NeuroRx. 2006 Jan;3(1):69-81. doi: 10.1016/j.nurx.2005.12.006. PMID 16490414
- [Background] Coric V, Taskiran S, Pittenger C, Wasylink S, Mathalon DH, Valentine G, Saksa J, Wu YT, Gueorguieva R, Sanacora G, Malison RT, Krystal JH. Riluzole augmentation in treatment-resistant obsessive-compulsive disorder: an open-label trial. Biol Psychiatry. 2005 Sep 1;58(5):424-8. doi: 10.1016/j.biopsych.2005.04.043. PMID 15993857
- [Background] Pittenger C, Bloch MH, Williams K. Glutamate abnormalities in obsessive compulsive disorder: neurobiology, pathophysiology, and treatment. Pharmacol Ther. 2011 Dec;132(3):314-32. doi: 10.1016/j.pharmthera.2011.09.006. Epub 2011 Sep 22. PMID 21963369
- See also: Yale OCD Research Clinic site — http://psychiatry.yale.edu/ocd/
- See also: Related Info — http://psychiatry.yale.edu/ocd/

RESULTS

PARTICIPANT FLOW:
Groups:
- N-Acetylcysteine: Patients randomized to this arm will receive N-Acetylcysteine augmentation, at a standard dose titrated to 3000 mg within the first week, in addition to the medication regimen they are on at enrollment
  N-Acetylcysteine : 3000 mg by mouth PO (1200 mg AM, 1800 mg PM), 12 weeks
- Placebo: Patients randomized to this arm will receive placebo, formulated to be indistinguishable from N-Acetylcysteine, in addition to the medication regimen they are on at study enrollment.
  placebo : placebo, 2 capsules PO AM, 3 capsules PO PM, 12 weeks
Period: Overall Study
Arm/Group | N-Acetylcysteine | Placebo
Started | 5 | 5
Received Allocated Intervention | 3 | 4
Completed | 3 | 3
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive-Compulsive Scale (Y-BOCS)at Baseline
Description: The Y-BOCS is a 10 item clinician-rated scale used to both determine the severity of OCD and to monitor symptom improvement throughout the course of the study. The Y-BOCS, specifically measures the severity of symptoms of obsessive-compulsive disorder without being biased towards the type of obsessions or compulsions present. The scale includes questions about the amount of time spent on, how much impairment or distress experienced from, and how much resistance and control over these obsessive thoughts and compulsions.
  Each item is rated from 0 ("no symptoms") to 4 ("extreme symptoms") and yields a total possible score range from 0 to 40, with the following ranges indicating degree of severity:
  0-7 = sub-clinical 8-15 = mild 16-23 = moderate 24-31 = severe 32-40 = extreme
  In this study, baseline ratings are compared to those of week 12 to produce a "percent of change" with positive percentages indicating a decrease in symptom severity.
Time Frame: Baseline
Population: Participants who completed the intervention were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 30.3 (5.7) | 28.6 (5.0)

2. Secondary Outcome: The Hamilton Depression Inventory (HAM-D)at Baseline
Description: The Hamilton Rating Scale for Depression is a multiple item (traditionally 17) assessment used to provide an indication of depression and as a guide to evaluate recovery. The clinician-rated assessment is designed for adults and is used to rate the severity of patient depression by asking about mood, feelings of guilt, insomnia, agitation, weight change, suicidal ideation, and somatic symptoms. The scale also allows the clinician to assess the patient's level of retardation, and insight into their depression.
  In this study, the HAM-D17 (17 items scored) was used to obtain depression severity ratings with a maximum possible score of 52. Baseline ratings are compared to those of week 12 to produce a "percentage of change", where positive values indicate a decrease in depressive severity/symptoms. Maximum score is a 52.
  Ranges
  0-7 = Normal 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression
  ≥23 = Very Severe Depression
Time Frame: Baseline
Population: Participants that completed the study were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 17.3 (2.3) | 8.7 (10.2)

3. Primary Outcome: Yale-Brown Obsessive-Compulsive Scale (Y-BOCS)at 12 Weeks
Description: as for outcome 1
Time Frame: 12 Weeks
Population: Participants who completed the intervention were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 30.6 (7.6) | 28.7 (1.6)

4. Secondary Outcome: The Hamilton Depression Inventory (HAM-D)at 12 Weeks
Description: as for outcome 2
Time Frame: 12 weeks
Population: Participants that completed the study were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 12.1 (8.2) | 7.0 (6.6)

ADVERSE EVENTS:
Arm/Group | N-Acetylcysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes